CLINICAL TRIAL: NCT03440463
Title: Alcohol Health Education With Personalized Feedback Boosters
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abby Braitman (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Abby Braitman, Research Assistant Professor, Old Dominion University
Organization: Old Dominion University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-221; K01AA023849 (NIH)
Record Dates: First submitted 2018-02-14; First posted 2018-02-22 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: College Student Drinking
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Who Masked: Participant
Masking Description: The intervention is an online program, not an individual, so masking is not necessary. Similarly, the same online survey is deployed in all follow-up assessments regardless of condition, and data are not collected by individuals, so masking is not necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention-only Control (Placebo Comparator): Participants navigate through e-checkup to go, the well-established alcohol intervention. Their email 2 weeks later contains only a reminder to participate in follow-up surveys.
  Interventions: Behavioral: e-checkup to go
- Intervention plus Norms-only booster (Experimental): Participants navigate through e-checkup to go, the well-established alcohol intervention. Their email 2 weeks later contains a reminder to participate in follow-up surveys, plus personalized feedback based on participant reported perceived alcohol norms, actual alcohol norms, and their own use.
  Interventions: Behavioral: e-checkup to go; Behavioral: Norms-only booster
- Intervention plus Norms-plus-Strategies booster (Experimental): Participants navigate through e-checkup to go, the well-established alcohol intervention. Their email 2 weeks later contains a reminder to participate in follow-up surveys, plus personalized feedback based on participant reported perceived alcohol norms, actual alcohol norms, and their own use. It also includes reported harm reduction strategies, and other strategies they might consider.
  Interventions: Behavioral: e-checkup to go; Behavioral: Norms-plus-Strategies booster

INTERVENTIONS:
Behavioral: e-checkup to go — The e-checkup to go substance program is designed to motivate individuals to reduce their consumption using personalized information about their own use and risk factors. The program is a combination of several components including alcohol education, personalized feedback, attitude-focused strategies, and skills training. It is self-guided and requires no face-to-face time with an administrator. It provides tailored feedback regarding quantity and frequency of alcohol use, normative comparisons, physical health information, amount and percent of income spent on alcohol, negative consequences feedback, explanation and advice for how to reach their goals, and resources.
Behavioral: Norms-only booster — Booster emails will contain normative feedback indicating average consumption for students at the same institution by sex, their perceptions of student drinkers at the same institution, their own reported consumption, and how they compare.
  Arms: Intervention plus Norms-only booster
Behavioral: Norms-plus-Strategies booster — Booster emails will contain normative feedback indicating average consumption for students at the same institution by sex, their perceptions of student drinkers at the same institution, their own reported consumption, and how they compare. These booster emails will also contain reminders of strategies they can use to protect themselves from alcohol-related harm, both ones they've reported using in the past and others they might consider using in the future.
  Arms: Intervention plus Norms-plus-Strategies booster

SUMMARY:
Heavy episodic alcohol use within the college student population is widespread, creating problems for student drinkers, their peers, and their institutions. Negative consequences from heavy alcohol use can be mild (e.g., hangovers, missed classes), to severe (e.g., assault, even death). Although online interventions targeting college student drinking reduce alcohol consumption and associated problems, they are not as effective as in-person interventions. Online interventions are cost-effective, offer privacy, reduce stigma, and may reach individuals who would otherwise not receive treatment.

In a recently completed randomized, controlled trial, an emailed booster with personalized feedback improved the efficacy of a popular online intervention (Braitman & Henson, 2016). Although promising, the booster incorporated in the study needs further empirical refinement. In addition, the intervention originally tested (Alcohol 101 Plus) is no longer widely available.

The current project seeks to build on past progress by further developing and refining the booster. In addition, it examines the utility of the booster after a different, widely-used, empirically-supported online intervention (e-checkup to go). e-checkup to go directly provides personalized normative feedback, but not protective strategies, the two components of the examined booster. Hence, the current study compares the reinforcing content (normative feedback) to the combination of reinforcing and novel content (norms PLUS protective strategies). There are 3 conditions: all participants receive the initial online intervention targeting college drinking. Condition 1 does not receive a booster email. Condition 2 receives an emailed booster with normative feedback only. Condition 3 receives an emailed booster with normative feedback plus protective strategies. The aims of the current study are as follows:

Aim 1: Examine if novel feedback in the form of protective strategies enhances the reinforcing normative feedback received via booster email (i.e., a comparison of reinforcing normative feedback only versus reinforcing normative feedback plus novel protective strategy feedback).

Aim 2: Examine previously identified potential moderators and mediators of reductions in alcohol use and related problems.

DETAILED DESCRIPTION:
Heavy episodic alcohol use within the college student population is widespread, creating problems for student drinkers, their peers, and their institutions. Negative consequences from frequent or heavy alcohol use can be mild (e.g., hangovers, missed classes), moderate (e.g., poor grades, damaged relationships), or severe (e.g., assault, even death). Given the potentially dangerous consequences, reducing alcohol use and associated problems is a major health priority. Although online interventions targeting college student drinking reduce alcohol consumption and associated problems, they are not as effective as in-person interventions. The benefits of online interventions include cost-effectiveness and ease of administration, plus they offer privacy, reduce stigma, and may reach individuals who would otherwise not receive treatment.

Although post-intervention boosters have been shown to be effective for individuals seeking treatment for alcohol-related injuries in emergency medical settings, limited studies have investigated the efficacy of boosters for college students who have received alcohol interventions. In a recently completed randomized, controlled trial, an emailed booster with personalized feedback improved the efficacy of a popular online intervention, while at the same time maintaining low cost and easy dissemination (Braitman & Henson, 2016). Although promising, the booster incorporated in the study needs further empirical refinement. In addition, the intervention originally tested (Alcohol 101 Plus) is no longer widely available.

The current project seeks to build on past progress reducing the gap between online and more efficacious in-person interventions. The current study further develops and refines the booster to identify optimal administration for maximum efficacy. In addition, it examines the utility of the booster after a different, widely-used, empirically-supported online intervention (e-checkup to go). The new intervention (e-checkup to go) directly provides personalized normative feedback, but not protective strategies, the two components of the examined booster. Hence, the current study compares the reinforcing content (personalized normative feedback) to the combination of reinforcing and enhancing/novel content (norms PLUS protective strategies). This addresses a major question of the relatively new booster literature for college drinking regarding if reinforcing content is sufficient to boost efficacy versus if novel information is an important supplementary component. There are 3 conditions: all participants receive the initial online intervention targeting college drinking. Condition 1 does not receive a booster email. Condition 2 receives an emailed booster with normative feedback only. Condition 3 receives an emailed booster with normative feedback plus protective strategies feedback. The booster content of tailored norms alone (reinforcing content) may alone be efficacious, or receiving tailored norms and strategies students can use to reduce consumption and related harm (protective behavioral strategies; novel content) may enhance the effect.

Thus, the aims of the current study are as follows:

Aim 1: Examine if novel feedback in the form of protective strategies enhances the reinforcing tailored normative feedback received via booster email (i.e., a comparison of reinforcing normative feedback only versus reinforcing normative feedback plus novel protective strategy feedback).

Hypothesis 1a: Both groups receiving emailed feedback will reduce drinking and alcohol-related problems as compared to the intervention-only control condition.

Hypothesis 1b: Reductions in drinking and problems will be stronger for those who receive emails with novel protective strategy feedback rather than reinforcing norms alone.

Aim 2: Examine previously identified potential moderators and mediators of reductions in alcohol use and related problems (i.e., gender, norms, strategies).

ELIGIBILITY:
Inclusion Criteria:

* Current college students at the sponsor institution at the time of enrollment
* Between the ages of 18 and 24
* Consumed at least standard drink of alcohol in the past 2 weeks

Exclusion Criteria:

* Under age of 18
* Over age of 24
* Not a college student
* Did not drink alcohol in the past 2 weeks

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 528 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby L Braitman, Ph.D., Principal Investigator — Old Dominion University
Locations (1):
- Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Braitman AL, Strowger M, Lau-Barraco C, Shipley JL, Kelley ML, Carey KB. Examining the added value of harm reduction strategies to emailed boosters to extend the effects of online interventions for college drinkers. Psychol Addict Behav. 2022 Sep;36(6):635-647. doi: 10.1037/adb0000755. Epub 2021 Jun 3. PMID 34081487

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Plus Norms-plus-Strategies Booster: Participants navigate through e-checkup to go, the well-established alcohol intervention. Their email 2 weeks later contains a reminder to participate in follow-up surveys, plus personalized feedback based on participant reported perceived alcohol norms, actual alcohol norms, and their own use. It also includes reported harm reduction strategies, and other strategies they might consider.
  e-checkup to go: The e-checkup to go program is designed to motivate individuals to reduce their consumption using personalized information about their own use and risk factors. The program is a combination of several components including alcohol education, personalized feedback, attitude-focused strategies, and skills training. It is self-guided and provides tailored feedback regarding quantity and frequency of alcohol use, normative comparisons, physical health information, amount and percent of income spent on alcohol, negative consequences feedback, explanation and advice for how to reach their goals, and resources.
  Norms-plus-Strategies booster: Booster emails contain normative feedback indicating average consumption for students at the same institution by sex, their perceptions of student drinkers at the same institution, and their own reported consumption. These emails also contain reminders of strategies they can use to protect themselves from alcohol-related harm, both ones they've reported using in the past and others they might consider using in the future.
Period: Baseline
Arm/Group | Intervention-only Control | Intervention Plus Norms-only Booster | Intervention Plus Norms-plus-Strategies Booster
Started | 201 | 163 | 164
Completed | 201 | 163 | 164
Not Completed | 0 | 0 | 0
Period: 1-month Follow-up
Arm/Group | Intervention-only Control | Intervention Plus Norms-only Booster | Intervention Plus Norms-plus-Strategies Booster
Started | 201 | 163 | 164
Completed | 134 | 113 | 107
Not Completed | 67 | 50 | 57
Period: 3-month Follow-up
Arm/Group | Intervention-only Control | Intervention Plus Norms-only Booster | Intervention Plus Norms-plus-Strategies Booster
Started | 201 | 163 | 164
Completed | 117 | 89 | 96
Not Completed | 84 | 74 | 68

BASELINE CHARACTERISTICS:
Population: Participants were students enrolled at a large, southeastern public university. To be eligible, participants must have been between the ages of 18-24, and consumed at least one alcoholic beverage in the previous 2 weeks.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention-only Control | Intervention Plus Norms-only Booster | Intervention Plus Norms-plus-Strategies Booster | Total
Number analyzed (Participants) | 201 | 163 | 164 | 528
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.80 (1.66) | 19.75 (1.53) | 20.02 (1.74) | 19.85 (1.65)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Participants were asked their gender with the response options of male, female, or other.
  Participants
    Male | 51 | 47 | 51 | 149
    Female | 150 | 115 | 113 | 378
    Other | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Asked via survey at baseline.
  Participants
    Hispanic or Latino | 176 | 146 | 145 | 467
    Not Hispanic or Latino | 25 | 17 | 16 | 58
    Unknown or Not Reported | 0 | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Asked via survey at baseline. Paricipants could select as many categories as they identified with, and this was recoded as "multiple races"
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 17 | 7 | 9 | 33
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 80 | 76 | 77 | 233
    White | 67 | 50 | 49 | 166
    More than one race | 20 | 25 | 18 | 63
    Unknown or Not Reported | 17 | 5 | 11 | 33
Drinks per typical week (quantity) [Mean (Standard Deviation); unit: drinks per week] | 8.18 (8.41) | 6.72 (7.14) | 8.05 (10.32) | 7.69 (8.71)
Drinking days per typical week (frequency) [Mean (Standard Deviation); unit: drinking days per week] | 2.24 (1.25) | 1.96 (1.13) | 2.23 (1.32) | 2.15 (1.24)
Highest drinking occasion in a typical week (peak) [Mean (Standard Deviation); unit: drinks per day] | 4.01 (2.98) | 3.48 (2.55) | 3.71 (3.20) | 3.76 (2.93)
Alcohol-related consequences (problems) [Mean (Standard Deviation); unit: score on a scale] — Assessed via the "Young Adult Alcohol Consequences Questionnaire" (Read et al., 2006). Participants indicate if they experienced an alcohol-related problem with a yes (=1) or no (=0). Scores are created by summing across all 48 items (range 0 to 48), where higher scores indicate experiencing more alcohol-related consequences/problems.
  Read, J. P., Kahler, C. W., Strong, D. R., & Colder, C. R. (2006). Development and preliminary validation of the young adult alcohol consequences questionnaire. Journal of Studies on Alcohol, 67, 169-177. doi:10.15288/jsa.2006.67.169
  score on a scale | 6.21 (6.59) | 6.07 (7.05) | 6.28 (7.17) | 6.19 (6.91)

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption at 3 Months Post-intervention
Description: Participant self-reported number of standard drinks consumed by participant in a typical week.
Time Frame: Past 30 days (3 months post-intervention)
Population: Participants who completed the follow-up survey 3 months post-intervention.
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Intervention-only Control | Intervention Plus Norms-only Booster | Intervention Plus Norms-plus-Strategies Booster
Number analyzed (Participants) | 117 | 89 | 96
drinks per week | 4.08 (5.81) | 4.15 (5.71) | 4.89 (7.68)

2. Secondary Outcome: Alcohol-related Consequences 3 Months Post-intervention
Description: Assessed via the "Young Adult Alcohol Consequences Questionnaire" (Read et al., 2006). Participants indicate if they experienced an alcohol-related problem with a yes (=1) or no (=0). Scores are created by summing across all 48 items (range 0 to 48), where higher scores indicate experiencing more alcohol-related consequences/problems.
  Read, J. P., Kahler, C. W., Strong, D. R., & Colder, C. R. (2006). Development and preliminary validation of the young adult alcohol consequences questionnaire. Journal of Studies on Alcohol, 67, 169-177. doi:10.15288/jsa.2006.67.169
Time Frame: Past 30 days (3 months post-intervention)
Population: Participants who completed the follow-up survey 3 months post-intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention-only Control | Intervention Plus Norms-only Booster | Intervention Plus Norms-plus-Strategies Booster
Number analyzed (Participants) | 117 | 89 | 96
score on a scale | 3.27 (5.68) | 2.37 (3.73) | 2.67 (4.11)

ADVERSE EVENTS:
Time Frame: 3 months post-intervention
Arm/Group | Intervention-only Control | Intervention Plus Norms-only Booster | Intervention Plus Norms-plus-Strategies Booster
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/163 | 0/164
Serious Adverse Events (participants affected / at risk) | 0/201 | 0/163 | 0/164
Other Adverse Events (participants affected / at risk) | 0/201 | 0/163 | 0/164

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT03440463/Prot_000.pdf
  • Informed Consent Form (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03440463/ICF_001.pdf